CLINICAL TRIAL: NCT05970497
Title: A Phase 1/2, Open-Label, Multi-Center, Dose Escalation and Expansion Study of KB707 in Subjects With Locally Advanced or Metastatic Solid Tumor Malignancies
Brief Title: A Study Assessing KB707 for the Treatment of Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Krystal Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KB707-01
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Cancer; Melanoma Stage III; Melanoma Stage IV; Cutaneous Melanoma
Keywords: Krystal Biotech; cancer; melanoma
MeSH Terms: conditions — Neoplasms; Melanoma | interventions — Opdualag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohorts 1 through 4 (Experimental): Dose escalation and expansion cohorts: KB707 monotherapy in subjects with solid tumors.
  Interventions: Biological: KB707
- Cohort 5 (Experimental): Dose expansion cohort: KB707 administered in combination with Opdualag in approximately 100 subjects with advanced melanoma.
  Interventions: Biological: KB707; Drug: Opdualag
- Cohort 6 (Experimental): Dose expansion cohort: KB707 administered in combination with Keytruda in approximately 100 subjects with advanced melanoma.
  Interventions: Biological: KB707; Drug: KEYTRUDA ®( Pembrolizumab)

INTERVENTIONS:
Biological: KB707 — Genetically modified herpes simplex type 1 virus
Drug: Opdualag — Dual immunotherapy (PD-1 and LAG-3 immune checkpoint inhibitors)
  Arms: Cohort 5
Drug: KEYTRUDA ®( Pembrolizumab) — Immunotherapy (PD-1 immune checkpoint inhibitor)
  Arms: Cohort 6

SUMMARY:
KB707-01 is a Phase 1/2, open-label, multicenter, dose escalation and expansion study. The study will evaluate the safety and tolerability of KB707 in adults with locally advanced or metastatic solid tumors who have progressed on standard of care therapy, cannot tolerate standard of care therapy, refused standard of care therapy, or for whom there is no standard of care therapy as well as the safety, tolerability, preliminary efficacy, and immunologic effect of KB707 administered in combination with Opdualag to subjects with unresectable or metastatic melanoma.

Subjects in dose escalation (Cohorts 1 through 3) and dose expansion (Cohort 4) will receive intratumoral injections of KB707 approximately every three weeks. Cohorts 1 through 4 are closed to new enrollment. Dose expansion Cohort 5 and Cohort 6 will evaluate subjects with advanced melanoma. Subjects in Cohort 5 will receive intratumoral injections of KB707 biweekly (q2w), delivered in combination with Opdualag (dosed every q4w per prescribing information). Subjects in Cohort 6 will receive intratumoral injections of KB707 biweekly (q2w), delivered in combination with Keytruda (dosed every q6w per prescribing information). All subjects will be treated until disease progression, death, unacceptable toxicity, symptomatic deterioration, achievement of maximal response, subject choice, Investigator decision to discontinue treatment, or the Sponsor determines to terminate the study.

DETAILED DESCRIPTION:
KB707 is a genetically modified herpes simplex type 1 virus that is designed to stimulate an anti-tumor immune response through the production of cytokines. This is a first-in-human (FIH) clinical study to evaluate the safety and tolerability and preliminary efficacy of KB707 in adult subjects with advanced and/or refractory solid tumors, including advanced melanoma. The study will include a dose escalation portion for single agent KB707 and an expansion portion to further evaluate single agent KB707 at a dose determined by preliminary data in the dose escalation phase as well as combination therapy of KB707 with immune checkpoint inhibitor therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Life expectancy >12 weeks
* ECOG performance status of 0 or 1
* Have measurable disease per RECIST v1.1 at Screening
* Cohorts 1-4 only: Histologically confirmed diagnosis of a locally advanced or metastatic solid tumor and the individual has progressed on standard of care therapy, cannot tolerate standard of care therapy, refused standard of care therapy, or there is no standard of care therapy.
* Cohorts 5 and 6 only: Histologically confirmed stage III (unresectable) or stage IV melanoma, as per American Joint Committee on Cancer (AJCC) staging system (8th edition; AJCC 2017) and

  1. Subject has previously failed one prior anti-PD-1/PD-L1 treatment (as monotherapy or in combination with other checkpoint inhibitors such as anti-LAG-3 or anti-CTLA-4); and
  2. If proto-oncogene B-Raf (BRAF) V600 mutation-positive, subject previously failed a BRAF inhibitor or BRAF inhibitor in combination with mitogen-activated extracellular signal-regulated kinase (MEK) inhibitor
* Cohort 5 only: Age 12 years or older at the time of informed consent
* Cohort 6 only: Age 18 years or older at the time of informed consent

Key Exclusion Criteria:

* Prior surgery or radiation therapy must be fully recovered, including all radiation -related toxicities and subject does not require systemic corticosteroids
* The subject is pregnant, nursing, or plans to become pregnant during study treatment and through three months after the last dose of KB707
* Have known history of positive human immunodeficiency virus (HIV 1/2)
* Cohorts 5 and 6 only:

  1. Subject has a known additional malignancy that is progressing or requires active treatment.
  2. Subject has uveal/ocular melanoma.
  3. The subject has active brain metastases or leptomeningeal metastases
  4. Subject has received more than 2 lines of systemic therapy for unresectable or metastatic melanoma
  5. Prior anti-LAG-3 and/or anti-PD-1 therapy was intolerable and required discontinuation of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of adverse events (AEs) | up to 36 months
  Percentage of subjects with adverse events (AEs)
Percentage of serious adverse events (SAEs) | up to 36 months
  Percentage of subjects with serious adverse events (SAEs)

SECONDARY OUTCOMES:
Maximum tolerated dose (MTD) | up to 36 months
  Assess whether the tested doses include the maximum tolerated dose (MTD) of KB707 based on the safety and response data collected during the dose escalation portion of the study
Percentage of overall response rate (ORR) | up to 36 months
  Percentage of ORR

CONTACTS AND LOCATIONS:
Overall Officials: David Chien, MD, Study Director — Senior Vice President of Clinical Development
Locations (15):
- United States (15):
  - UCLA Health, Los Angeles, California
  - Mission Dermatology Center, Rancho Santa Margarita, California
  - BRCR Global, Weston, Florida
  - IU Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Henry Ford Cancer Institute, Detroit, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Morristown Medical Center / Atlantic Health System, Morristown, New Jersey
  - Weill Cornell Medicine-New York-Presbyterian Hospital, New York, New York
  - Gabrail Cancer Center Research, Canton, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Renovatio Clinical - El Paso, El Paso, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Renovatio Clinical - The Woodlands, The Woodlands, Texas